CLINICAL TRIAL: NCT01211600
Title: Cesarean Randomized Control Trial Of Sutures vs. Staples (CROSS)
Brief Title: Cesarean Trial of Staples vs. Sutures
Acronym: CROSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Main Line Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10D.199
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cesarean Section; Wound Complications; Patient Satisfaction; Pain Measurement
Keywords: Staples; Sutures; Wound infections; Cosmesis; Aesthetic appearance of skin incision
MeSH Terms: conditions — Patient Satisfaction; Wound Infection | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Staples (Active Comparator): Interrupted Ethicon Staples
  Interventions: Other: Staples
- Suture (Active Comparator): Subcuticular continuous suture (4-0 Monocryl Plus on PS2 needle or 4-0 Vicryl Plus on FS2 or PS2 needle)
  Interventions: Other: Suture

INTERVENTIONS:
Other: Staples — Interrupted Ethicon Staples
  Other Names: Closure Technique
  Arms: Staples
Other: Suture — Subcuticular continuous suture (4-0 Monocryl Plus on PS2 needle or 4-0 Vicryl Plus on FS2 or PS2 needle)
  Other Names: Closure Technique
  Arms: Suture

SUMMARY:
To determine whether the rate of wound complications differs based on method of closure of skin incision (staples vs. suture) after cesarean delivery.

DETAILED DESCRIPTION:
Despite this large number of cesareans performed annually, there is a paucity of data to suggest which technique is superior for closure of the skin incision with regards to wound complications, including wound separation and infection. As the morbidity associated with a cesarean delivery is usually related to wound complications, especially infection, we feel that it is important to examine this outcome by comparing the current skin closure techniques: staples versus suture.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing cesarean delivery for pregnancy greater than 23 weeks gestation.

Exclusion Criteria:

* Poorly controlled diabetes (defined as ≥ 50% of fasting or 2 hour postprandial glucose levels > 95 and 120 respectively within the week prior to delivery),
* Vertical skin incisions
* Chronic steroid use
* Active lupus flare
* HIV/AIDS
* Current treatment for cancer or a history of radiation to the abdomen/pelvis
* Current treatment with immunosuppressant medications secondary to history of transplantation
* Emergency cesarean(precluding informed consent prior to surgery)
* Lack of access to a phone
* Allergy to suture or staple material

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2010-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Dhanya Mackeen, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Alderdice F, McKenna D, Dornan J. Techniques and materials for skin closure in caesarean section. Cochrane Database Syst Rev. 2003;(2):CD003577. doi: 10.1002/14651858.CD003577. PMID 12804476
- [Background] Basha SL, Rochon ML, Quinones JN, Coassolo KM, Rust OA, Smulian JC. Randomized controlled trial of wound complication rates of subcuticular suture vs staples for skin closure at cesarean delivery. Am J Obstet Gynecol. 2010 Sep;203(3):285.e1-8. doi: 10.1016/j.ajog.2010.07.011. PMID 20816153
- [Derived] Mackeen AD, Khalifeh A, Fleisher J, Han C, Leiby B, Berghella V. Pain Associated With Cesarean Delivery Skin Closure: A Randomized Controlled Trial. Obstet Gynecol. 2015 Oct;126(4):702-707. doi: 10.1097/AOG.0000000000001043. PMID 26348166
- [Derived] Mackeen AD, Khalifeh A, Fleisher J, Vogell A, Han C, Sendecki J, Pettker C, Leiby BE, Baxter JK, Sfakianaki A, Berghella V. Suture compared with staple skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1169-1175. doi: 10.1097/AOG.0000000000000227. PMID 24807325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suture | Staples
Started | 370 | 376
Completed | 370 | 376
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture | Staples | Total
Number analyzed (Participants) | 370 | 376 | 746
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 31.0 [26.9 to 35.4] | 31.0 [26.4 to 35.6] | 31.0 [26.6 to 35.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 376 | 746
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 158 | 167 | 325
  Caucasian | 162 | 154 | 316
  Hispanic | 19 | 24 | 43
  Asian | 16 | 22 | 38
  Other | 15 | 8 | 23
  Unknown | 0 | 1 | 1
Pregnancy History - Singleton Gestation [Count of Participants; unit: Participants] — Number of participants with singleton pregnancy
  Participants | 353 | 351 | 704
Number of Previous Cesareans [Count of Participants; unit: Participants] — Participants who had 0, 1, or more than one cesarean prior to study participation
  Participants
    0 Previous Cesareans | 180 | 177 | 357
    1 Previous Cesarean | 120 | 132 | 252
    More than 1 Previous Cesarean | 70 | 67 | 137
Term Gestation [Count of Participants; unit: Participants] — Number of participants at 37 weeks or greater gestation at time of participation.
  Participants | 317 | 329 | 646

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complications
Description: The primary outcome is to evaluate the rate of wound complications for patients undergoing cesarean whose skin incision is closed with staples versus with suture.
  Wound complications included infection, hematoma, seroma, and separation and readmission for wound complication.
Time Frame: Within 6 weeks of postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Participants
  Total patients with at least 1 wound complicatin | 18 | 40
  Infection | 9 | 14
  Hematoma | 2 | 4
  Seroma | 5 | 6
  Separation | 6 | 28
  Readmission for wound complication | 2 | 3

2. Secondary Outcome: Patient Scar Assessment Scale Scores for Evaluation of Cosmesis
Description: Patient evaluation of cosmesis of the cesarean incision based on closure method: staples vs sutures.
  Surgical scars were evaluated using Patient Scar Assessment Scale (PSAS). The PSAS evaluates six items: pain, itchiness, color, stiffness, thickness, and irregularity. Each item is scored on a 10-point scale comparing the patient's skin to normal skin, in which one represents normal skin. The score is summed, range 6-60. Lower scores indicate closer resemblance to normal skin and are superior.
Time Frame: Immediately postpartum and 4 - 8 weeks after intervention, up to 12 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suture | Staples
Number analyzed (Participants) | 286 | 291
score on a scale | 15 [10 to 25] | 20 [11 to 28]

3. Secondary Outcome: Patient Satisfaction With Closure Method and Scar Appearance
Description: Whether the patient's satisfaction with the incision differed based on closure method (staples vs sutures) using 10-point Likert scale on which 1 is completely dissatisfied and 10 is completely satisfied.
Time Frame: Immediately postpartum and 4 - 8 weeks after intervention, up to 12 weeks.
Population: Patient satisfaction data were available for 606 participants. Two participants in the Staples arm did not provide scores for scar appearance satisfaction. This is why we are representing 305 of the 307 subjects' responses to satisfaction of scar appearance.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Staples | Suture
Number analyzed (Participants) | 307 | 299
score on a scale
  Satisfaction with Closure Method | 9 [6 to 10] | 10 [9 to 10]
  Satisfaction with Scar Appearance: number analyzed (Participants) | 305 | 299
  Satisfaction with Scar Appearance | 9 [7 to 10] | 9 [8 to 10]

4. Secondary Outcome: Pain Perception
Description: Whether the patient's perception of pain associated with the incision differed based on closure method (staples vs sutures). Patients were asked to rate pain on a scale from 0 (no pain) to 10 (extreme pain) using a visual graph of facial expressions.
Time Frame: Immediately postpartum to time of discharge, which is typically 3-4 days post-cesarean
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
score on a scale
  Less than 24 hours | 3.5 [2.0 to 5.0] | 3.6 [2.2 to 5.0]
  24 - 47 hours | 4.3 [3.5 to 5.2] | 4.3 [3.4 to 5.2]
  48 - 72 hours | 4.3 [3.5 to 5.3] | 4.2 [3.3 to 5.1]
  Pain at time of Discharge | 3.5 [2.0 to 5.0] | 3.6 [2.2 to 5.0]

5. Secondary Outcome: Additional Provider Visits
Description: Mean number of visits per participant (All wound visits, number of visits for women who were diagnosed with wound complications, number of visits for women who were not diagnosed with a wound complication).
Time Frame: Within 6 weeks postpartum
Population: The number analyzed in the "Number of visits - diagnosed wound complication" and "Number of visits - no diagnosed wound complication" rows indicates the breakdown of subjects within each arm that did and did not have a diagnosed wound complication.
Measure: Mean (Full Range); unit: Number of Visits per participant
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Number of Visits per participant
  All wound visits | .9 [0 to 7] | 1.5 [0 to 7]
  Number of visits - diagnosed wound complication: number analyzed (Participants) | 18 | 40
  Number of visits - diagnosed wound complication | 2.7 [1 to 7] | 2.9 [1 to 7]
  Number of visits - no diagnosed wound complication: number analyzed (Participants) | 352 | 336
  Number of visits - no diagnosed wound complication | .8 [0 to 3] | 1.4 [0 to 6]

6. Secondary Outcome: Number of Participants With Primary Versus Repeat Cesarean
Description: Randomization stratum - BMI (over/under 30) and Cesarean (primary or repeat)
Time Frame: At randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Participants
  BMI 30 or greater - primary cesarean delivery | 109 | 106
  BMI 30 or greater - repeat cesarean delivery | 126 | 132
  BMI less than 30 - primary cesarean delivery | 71 | 71
  BMI less than 30 - repeat cesarean delivery | 64 | 67

7. Secondary Outcome: Intraoperative Trial Details - Duration of Operation and Skin Closure
Description: Duration of operation: skin incision to skin closure Duration of skin closure: fascial closure to skin closure
Time Frame: Time of Cesarean
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Minutes
  Duration of Operation | 58.5 [46.5 to 75] | 51 [40 to 65]
  Duration of Skin Closure | 15 [12 to 19] | 6 [4 to 9]

8. Secondary Outcome: Intraoperative Trial Details - Closure of Subcutaneous Tissue
Description: Number of participants requiring subcutaneous tissue closure
Time Frame: Time of Cesarean
Measure: Count of Participants; unit: Participants
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Participants | 201 | 202

9. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay (days)
Time Frame: Immediate postpartum.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Days | 4.4 [1 to 8] | 4.5 [3 to 14]

10. Secondary Outcome: Number of Participants That Received Anticoagulation Within 24 Hours
Description: Number of participants that received anticoagulation within 24 hours of procedure (preoperatively or postoperatively)
Time Frame: Within 24 hours postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Participants | 14 | 17

11. Secondary Outcome: Number of Participants Diagnosed With Endomyometritis
Description: Number of participants diagnosed with endomyometritis requiring antibiotics
Time Frame: Immediate postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
Participants | 11 | 7

12. Secondary Outcome: Change in Hemoglobin Pre-operatively to Post-operatively
Description: Median change in hemoglobin from preoperative value (g/dL) to post-operatively.
Time Frame: Up to 72 hours before and 24 hours after cesarean.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Suture | Staples
Number analyzed (Participants) | 370 | 376
g/dL | -1.8 [-2.5 to -1.2] | -1.8 [-2.5 to -1.1]

13. Secondary Outcome: Observer Evaluation of Cosmesis of the Cesarean Incision Based on Closure Method: Staples vs Sutures.
Description: Surgical scars were evaluated using Observer Scar Assessment Scale (OSAS). The OSAS evaluates five items: vascularity, pigmentation, thickness, relief, and pliability. Each item is scored on a 10-point scale comparing the patient's skin to normal skin, in which one represents normal skin. The score is summed, range 5-50. Lower scores indicate closer resemblance to normal skin and are superior.
Time Frame: Immediately postpartum and 4 - 8 weeks after intervention, up to 12 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suture | Staples
Number analyzed (Participants) | 137 | 138
score on a scale | 12 [9 to 15] | 13 [9 to 16]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of randomization to 30 days postpartum.
Arm/Group | Suture | Staples
All-Cause Mortality (participants affected / at risk) | 0/370 | 0/376
Serious Adverse Events (participants affected / at risk) | 0/370 | 0/376
Other Adverse Events (participants affected / at risk) | 18/370 | 40/376
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suture (N=370) | Staples (N=376)
Wound Complications (Skin and subcutaneous tissue disorders) | 18 (18) | 40 (40) — Wound complications are a known risk of both cesarean closure methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No